CLINICAL TRIAL: NCT06357598
Title: Preoperative Neoadjuvant Immunotherapy Combined With Chemotherapy for Newly Diagnosed Stage Ⅲ Unresectable Non-small Cell Lung Cancer: a Open-label, Single-arm Prospective Clinical Trial
Brief Title: Preoperative Neoadjuvant Immunotherapy Combined With Chemotherapy for Stage Ⅲ Unresectable Non-small Cell Lung Cancer
Acronym: PILOT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jiaowenjie, Professor, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2023-95
Record Dates: First submitted 2024-03-28; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Non-small-cell Lung Cancer (NSCLC)
Keywords: Non-small-cell Lung Cancer (NSCLC); Immunotherapy; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; spartalizumab; Pemetrexed; Antineoplastic Agents; Carboplatin; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Participants receive 2-4 cycles of Tislelizumab combined with chemotherapy treatment during preoperative period, every 3 weeks for 4 cycles at most.
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed (Non-squamous NSCLC) or Nab-paclitaxel(Squamous NSCLC); Drug: Carboplatin or Cisplatin; Procedure: Surgery

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200mg, ivgtt, day 1 of each 21-day cycle, neoadjuvant therapy : 2-4 cycles; Adjuvant therapy: 16cycles at most.
  Other Names: PD-1 antibody
Drug: Pemetrexed (Non-squamous NSCLC) or Nab-paclitaxel(Squamous NSCLC) — Pemetrexed: 500 mg/m^2, ivgtt, day 1 of each 21-day cycle, 2-4 cycles. Nab-paclitaxel: 260mg/m^2, ivgtt, day 1 of each 21-day cycle, 2-4 cycles.
  Other Names: chemotherapeutic drug
Drug: Carboplatin or Cisplatin — Carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 5 ivgtt on day 1 of each 21-day cycle for 2-4 cycles.
  Cisplatin: 75 mg/m^2, ivgtt, day 1 of each 21-day cycle, 2-4 cycles.
  Other Names: chemotherapeutic drug
Procedure: Surgery — Surgery must be done within the 4th-6th week from day 1 the last cycle of neoadjuvant treatment.

SUMMARY:
Explorative study, which evaluates the effect of Tislelizumab combined with chemotherapy in neoadjuvant treatment of stage Ⅲ unresectable non-small-cell lung carcinoma.

DETAILED DESCRIPTION:
This is a open-label, single-arm prospective clinical trial to evaluate the efficacy and safety of Tislelizumab combined with chemotherapy in neoadjuvant treatment of newly diagnosed stage Ⅲ unresectable non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age :18 Years to 75 Years;
2. ECOG physical score status of 0 or 1 points;
3. Expected survival time ≥ 6 months;
4. According to the eighth edition of the AJCC/UICC TNM staging system, patients were pathological diagnosed with Stage III NSCLC and had one of the following conditions: 1) A complete resection (R0) would not be possible, based on evaluation within a multidisciplinary team, including an experienced thoracic surgeon; 2) Multiple ipsilateral mediastinal lymph nodes metastasized into large masses or multistation metastases (IIIA: T1-2N2 or IIIB: T3-4N2); 3) Contralateral hilar or mediastinal lymph nodes, or ipsilateral or contralateral scalene or supraclavicular lymph nodes metastasis (IIIB: T1-2N3; IIIC: T3-4N3); 4) The lesion invaded the heart, aorta, or esophagus (IIIA: T4N0-1).
5. EGFR mutation or ALK mutation was negative;
6. Patients with at least one evaluable or measurable lesions as per RECIST version 1.1;
7. Patients were newly diagnosed with non-small cell lung cancer, without radiotherapy, chemotherapy, surgery or molecule-targeted treatment.
8. Patients must have enough cardiopulmonary function for the expected pulmonary resections for lung cancer.
9. The main organ function meets the following criteria:1) Blood routine:a. ANC ≥ 1.5×109/L; b. PLT ≥ 100×109/L; c. HB ≥ 90 g/L; 2) Blood biochemistry:TBIL ≤ 1.5×ULN;ALT、AST≤ 2.5×ULN;sCr≤1.5×ULN; 3) Blood coagulation: INR≤1.5×ULN and APTT≤1.5×ULN，endogenous creatinine clearance rate≥45ml/min(Cockcroft-Gault formula);
10. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 3 months post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 3 months post the last administration of study drug;
11. Patient has to voluntarily join the study and sign the Informed Consent Form for the study.

Exclusion Criteria:

1. Patients with autoimmune disease, or a history of autoimmune disease within 2 years prior to the first use of the study drug including but not limited to the following: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism which can be included after hormone replacement therapy; Subjects with childhood asthma have been completely alleviated and without any intervention or vitiligo in adulthood can be included;
2. Subjects with congenital or acquired immunodeficiency such as HIV infection, active hepatitis B (HBV DNA ≥ 2000 IU/mL), hepatitis C (hepatitis C antibody is positive);
3. Subjects with a condition requiring other immunosuppressive medications before 7 days of study drug administration firstly, not including inhaled corticosteroids or physiological doses of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents);
4. Has received a live vaccine within 4 weeks of planned start of study therapy;
5. Other malignancies have been diagnosed within 5 years prior to the first use of the study drug (excluding skin basal cell carcinoma that has been cured, skin squamous cell carcinoma, and / or carcinoma in situ that has undergone radical resection);
6. Patients with a current or history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiologic pneumonia, drug-induced pneumonia and severe impairment of lung function;
7. Patients with serious or uncontrollable systemic diseases, such as:

   Patients with hypertension that is difficult to control (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg); Patients with myocardial ischemia and myocardial infarction above class II (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms);
8. Severe infection within 4 weeks before the first administration (such as intravenous drip of antibiotics, antifungal drugs or antiviral drugs), or fever of unknown origin (> 38.5 ℃) within 4 weeks before the first administration;
9. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
10. Pregnant or nursing women;
11. Patients with a history of hypersensitivity to any of the study drugs, similar drugs, or excipients;
12. Participated in other clinical trials within 4 weeks;
13. Patients has received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulator or synergistically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137);
14. The investigator believes that there are any conditions that may damage the subject or result in the subject being unable to meet or perform the research request.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | 1 month after surgery
  R0 Resection Rate: The pathological results will showed that the incision margin was negative and no residual cancer cells were found under the microscope.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Pre-operation
  Objective Response Rate (ORR): defined as the proportion of patients whose tumor size shrinks to predefined values，which including cases of CR and PR. Objective tumor response will be assessed using RECIST 1.1. Subjects must have measurable tumor lesions at baseline, and the response evaluation criteria are classified as complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to RECIST 1.1.
Resectability Rate | Pre-operation
  Resectability Rate is defined as the percentage of patients who were able to undergo surgery after neoadjuvant therapy.
Major Pathological Response (MPR) Rate | 1 month after surgery
  Major Pathological Response (MPR) Rate: defined as ≤ 10% of residual tumor cells in the surgically resected tumor specimen and sampled regional lymph nodes after neoadjuvant treatment.
Rate of grade 3 and higher grade treatment-related adverse events | From date of treatment allocation until surgery or within 30 days after last dose of preoperative treatment
  Adverse events will be evaluated and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).
Progression-Free Survival (PFS) | Up to 12 months
  Progression-Free Survival (PFS): defined as the time from the first dose until the date of first documented progression or date of death from any cause, whichever came first.

OTHER OUTCOMES:
Pathological Complete Response (pCR) Rate | 1 month after surgery
  Pathological Complete Response (pCR) Rate: no residual tumor cells in the surgically resected tumor specimen and all sampled regional lymph nodes after neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Jiao, PhD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No